CLINICAL TRIAL: NCT06481332
Title: Diagnostic Characterization and Evolution of "Triple Negative" Thrombocytosis
Brief Title: Diagnostic Characterization and Evolution of "Triple Negative" Thrombocytosis (CASTETTE)
Acronym: CASTETTE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0135 - CASTETTE
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-04

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of Event free survival in patients with triple-negative thrombocytosis

DETAILED DESCRIPTION:
Patients with non-reactive thrombocytosis, explored at least by bone marrow biopsy and NGS panel will be included. Clinical and biological characteristics as well as evolution will be recorded retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non reactive thrombocytosis for at least 6 months
* availability of bone marrow biopsy and NGS panel

Exclusion Criteria:

* Unable to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients followed by hematologists of the French Intergroup of MPN
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement